CLINICAL TRIAL: NCT05445570
Title: Non-invasive Identification of Colorectal Cancer and Adenomas in Early Stages
Acronym: NICE
Status: Completed | Type: Observational
Sponsor: Venn Biosciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: NICE-001
Record Dates: First submitted 2022-04-21; First posted 2022-07-06 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample will be collected at baseline for all subjects. blood sample will be collected at follow-up for a subgroup of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Non-Interventional — This is an observational, non interventional study

SUMMARY:
The NICE study is a prospective, multi-site study to train and validate a blood-based, glycoproteomic test for the early detection of advanced adenoma and colorectal cancer by collecting blood samples and associated relevant clinical information from average-risk participants who undergo routine screening colonoscopy as well as participants undergoing colonoscopy for surveillance or diagnostic indications

DETAILED DESCRIPTION:
InterVenn is using its glycoprotein profiling technology platform that couples high-resolution liquid chromatography (LC)-mass spectrometry (MS) with an artificial intelligence (AI), neural network (NN)-based high-throughput data processing software to identify patterns uniquely associated with colon adenoma and colon adenocarcinoma in order to detect (pre)cancerous events early. The purpose of this prospective multi-center observational study is to train and validate a blood-based, glycoproteomic test for the early detection of advanced adenoma and colorectal cancer by collecting blood samples and associated relevant clinical information from average-risk participants who undergo routine screening colonoscopy as well as participants undergoing colonoscopy for surveillance or diagnostic indications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 45-85.
2. Able to provide an informed consent and who understand and agree to all study procedures required
3. Subject is scheduled or will soon be scheduled to receive a colonoscopy as ordered by their doctor.

Exclusion Criteria:

1. Any active malignancy
2. Any other illness that in the opinion of the investigator, makes the subject not a good candidate for the study.

Ages: 45 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population comprises approximately 3000 subjects, male and female, between the ages of 45 and 85 who are scheduled for or will soon be scheduled for a screening, surveillance, or diagnostic colonoscopy.
Sampling Method: Probability Sample
Enrollment: 3002 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the InterVenn test | up to 90 days from baseline
  To determine the sensitivity of the InterVenn test
Specificity of the InterVenn test | up to 90 days from baseline
  To determine the specificity of the InterVenn test

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hommes, MD, Study Director — InterVenn Biosciences
Locations (12):
- United States (12):
  - East View Medical Research, LLD, Mobile, Alabama
  - Paragon Rx Clinical, Garden Grove, California
  - Paragon Rx Clinical, Santa Ana, California
  - Encore - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Encore - Nature Coast Clinical Research, Inverness, Florida
  - Encore - Westside Center for Clinical Research, Jacksonville, Florida
  - Encore Borland Groover, Jacksonville, Florida
  - Encore - St. Johns Center for Clinical Research, Saint Augustine, Florida
  - Combined Gastro Research, LLC, Lafayette, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Allied Health Clinical Research Organization, Freehold, New Jersey
  - Blue Ridge Medical Research, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- See also: Sponsor Website — https://intervenn.com/